CLINICAL TRIAL: NCT02447094
Title: Assessing the Impact of Care in A Telemedicine-based Stroke Network Using Patient-Centered Health Related Quality of Life Outcomes
Brief Title: Quality of Life After Stroke Using a Telemedicine-based Stroke Network
Acronym: STROKE TeleQOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Fred Rincon, Assistant Professor of Neurology and Neurosurgery, Thomas Jefferson University
Other Study IDs: 15D.044
Record Dates: First submitted 2015-05-09; First posted 2015-05-18 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Stroke
Keywords: ischemic; tPA; tele-medicine; robot; tele-stroke
MeSH Terms: conditions — Stroke; Ischemia | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed: AIS patients evaluated through RTP and who receive i.v. tPA
  Interventions: Drug: Alteplase
- Un-exposed: AIS patients evaluated through RTP and who do not receive i.v. tPA

INTERVENTIONS:
Drug: Alteplase — Intravenous (i.v.) tPA per the standard of care
  Other Names: Recombinant tissue plasminogen activator (tPA)
  Groups: Exposed

SUMMARY:
To study the effect of a telemedicine model of stroke care on patient-based outcomes.

DETAILED DESCRIPTION:
Approximately 750,000 patients suffer from ischemic stroke (AIS) annually in the United States. AIS is a a leading cause of long-term disability and the third-leading cause of mortality. Effective therapies exist to ameliorate the disability associated with AIS, but implementation of these therapies is time-sensitive. Currently, there is a shortage in health care professionals with expertise in the treatment of stroke and such expertise tends to be concentrated in large community-based or academic medical centers. To respond to this shortage, stroke networks are being organized in a "hub-and-spoke" model to facilitate the rapid delivery of time-sensitive interventions such as intravenous (i.v.) tissue plasminogen activator (tPA) or rapid evaluation for AIS. Some networks are also using telemedicine to facilitate this approach and bring the needed expertise via robotic tele-presence (RTP). Though the accuracy of stroke diagnosis and i.v. tPA utilization may be higher in RTP based networks, the impact of this model on patient's outcomes has been difficult to elucidate. To this end, meaningful validated outcome assessments are crucial to understand the impact of stroke interventions including telemedicine or RTP based networks. The objective of this study is to translate evidence-based practice of healthcare, patient-centered outcome assessments, and patient-family perceptions of delivery of care into meaningful data. This will aid in the validation of the role of interventions such as "hub-and-spoke" RTP based models in stroke care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected acute ischemic stroke (AIS)
* Age >17 years

Exclusion Criteria:

* Hemorrhagic strokes (ICH or SAH)
* Transient ischemic attacks (TIA)
* Trauma
* Inability to obtain informed consent
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research will be performed only in AIS patients who are routinely admitted to our "Hub" and participating "spoke" centers.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
HRQoL | 6 months
  Health Related Quality of Life

SECONDARY OUTCOMES:
mRS | 6 months
  Modified Rankin Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States